CLINICAL TRIAL: NCT05858450
Title: Investigating Uptake and Subsequent Health Outcomes Associated With Pfizer-BioNTech Bivalent COVID-19/Influenza Vaccine Concomitant Administration Using a Claims-based Real-world Data Source in the US
Brief Title: This Study Intends to Describe the Characteristics of Patients Given the Pfizer-BioNTech Bivalent mRNA COVID-19 Vaccine and Any Commercially Available Influenza Vaccines at the Same Time Versus at Different Times.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591061
Record Dates: First submitted 2023-05-11; First posted 2023-05-15 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Influenza, Human; COVID-19
MeSH Terms: conditions — Influenza, Human; COVID-19 | interventions — BNT162 Vaccine; Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Same day: Pfizer-BioNTech mRNA bivalent COVID and flu on the same day
  Interventions: Biological: Comirnaty; Biological: Quadrivalent Influenza Vaccine
- COVID alone: Pfizer-BioNTech bivalent COVID only
  Interventions: Biological: Comirnaty
- flu alone: influenza vaccine of any type only
  Interventions: Biological: Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Comirnaty — COMIRNATY is an active immunization to prevent COVID-19 caused by SARS-CoV-2 in individuals 12 years of age and older.
  Groups: COVID alone; Same day
Biological: Quadrivalent Influenza Vaccine — Quadrivalent Influenza Vaccine is a class of vaccines indicated for active immunization for the prevention of influenza disease caused by influenza A subtype viruses and type B viruses contained in the vaccines
  Groups: Same day; flu alone

SUMMARY:
This study intends to describe the characteristics of patients given the Pfizer-BioNTech bivalent mRNA COVID-19 vaccine and any commercially available influenza vaccines at the same time versus at different times.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Optum claims database as of 31 August 2022 (date bivalent authorized).
* Has a Pfizer-BioNTech mRNA bivalent COVID-19 or influenza vaccine (any type) between 31 August 2022 and 30 January 2023 (earliest vaccine is index date).
* Aged >=18 years on the index date
* 365 days of continuous enrolment prior to index date

Exclusion Criteria:

* Patients with a second dose of any type of bivalent mRNA COVID-19 or flu vaccine, disenrolled or died within 14 days following the first dose.
* Has prior COVID-19 diagnosis (U07.1, any setting, any position) within 90 days (per CDC guidance on length of time before receiving a vaccine) before and on index.
* Has influenza vaccine between 01 August -30 August 2022 (before study period).
* Has a COVID-19 or influenza diagnosis code in any setting within 14 days after index vaccination (excluded from all cohorts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults patients who were enrolled in the Optum Clinformatics Database as of 31 August 2022
Sampling Method: Non-Probability Sample
Enrollment: 3442996 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants (greater than or equal to [>=] 18 years) who were enrolled in the Optum Clinformatics Database as of 31 August 2022 and had received a Pfizer-BioNTech messenger ribonucleic acid (mRNA) bivalent COVID-19 vaccine and/or seasonal influenza/flu vaccine (SIV) anytime between 31 August 2022 and 30 January 2023 were included in this retrospective, observational study.
Pre-assignment Details: Outcome measures were compared using Cox Proportional Hazards models for the following exposure groups: comparison 1: co-administration of vaccines on the same day and COVID-19 vaccine alone, comparison 2: co-administration of vaccines on the same day (excluded participants with unknown/other region) and SIV alone.
Groups:
- Group 1a: Same Day COVID-19 Vaccine and SIV, 18-64 Years: Participants included in this group were aged 18-64 years, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine and SIV on the same day (co-administration) anytime between 31 August 2022 and 30 January 2023.
- Group 2a: COVID-19 Vaccine Alone, 18-64 Years: Participants included in this group were aged 18-64 years, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine alone any time between 31 August 2022 and 30 January 2023.
- Group 3a: SIV Alone, 18-64 Years: Participants included in this group were aged 18-64 years, who were enrolled in the Optum Clinformatics Database and received SIV alone any time between 31 August 2022 and 30 January 2023.
- Group 1b: Same Day COVID-19 Vaccine and SIV, >= 65 Years: Participants included in this group were aged 65 years and above, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine and SIV (enhanced) on the same day (co-administration) anytime between 31 August 2022 and 30 January 2023.
- Group 2b: COVID-19 Vaccine Alone, >=65 Years: Participants included in this group were aged 65 years and above, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine alone any time between 31 August 2022 and 30 January 2023.
- Group 3b: SIV Alone, >=65 Years: Participants included in this group were aged 65 years and above, who were enrolled in the Optum Clinformatics Database and received SIV (enhanced) alone any time between 31 August 2022 and 30 January 2023.
Period: Overall Study
Arm/Group | Group 1a: Same Day COVID-19 Vaccine and SIV, 18-64 Years | Group 2a: COVID-19 Vaccine Alone, 18-64 Years | Group 3a: SIV Alone, 18-64 Years | Group 1b: Same Day COVID-19 Vaccine and SIV, >= 65 Years | Group 2b: COVID-19 Vaccine Alone, >=65 Years | Group 3b: SIV Alone, >=65 Years
Started | 244900 | 143743 | 843860 | 382835 | 225680 | 1601978
Completed | 244900 | 143743 | 843860 | 382835 | 225680 | 1601978
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants whose data were observed in this retrospective observational study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1a: Same Day COVID-19 Vaccine and SIV, 18-64 Years | Group 2a: COVID-19 Vaccine Alone, 18-64 Years | Group 3a: SIV Alone, 18-64 Years | Group 1b: Same Day COVID-19 Vaccine and SIV, >= 65 Years | Group 2b: COVID-19 Vaccine Alone, >=65 Years | Group 3b: SIV Alone, >=65 Years | Total
Number analyzed (Participants) | 244900 | 143743 | 843860 | 382835 | 225680 | 1601978 | 3442996
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 244900 | 143743 | 843860 | 0 | 0 | 0 | 1232503
  65 years and above | 0 | 0 | 0 | 382835 | 225680 | 1601978 | 2210493
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 127108 | 78029 | 477067 | 208166 | 132345 | 939216 | 1961931
  Male | 117692 | 65655 | 366067 | 174651 | 93327 | 661737 | 1479129
  Unknown | 100 | 59 | 726 | 18 | 8 | 1025 | 1936
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/ethnicity data was not available.
  Participants
    Data not available | 244900 | 143743 | 843860 | 382835 | 225680 | 1601978 | 3442996

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All Cause Hospitalization Visits: 18-64 Years Old
Description: Hospitalization due to any cause is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility). To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs Flu (SIV) alone.
Time Frame: From Day 15 of vaccination till end of follow-up observation period, from 14-Sep-2022 through 14 February 2023 (approximately 5 months); data was extracted and observed in this retrospective study from 05-May-2023 to 12-May-2023 (8 days)
Population: All eligible participants whose data were observed in this study. This outcome measure presents reporting arms as planned based on the following: participants 18-64 years of age for both models: Model 1 (reporting arms included were co-administration of vaccines on the same day and COVID-19 alone), Model 2 (reporting arms included were co-administration of vaccines on the same day [excluded participants with unknown/other region] and SIV alone).
Measure: Count of Participants; unit: Participants
Groups:
- Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years: Participants aged 18-64 years, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine and SIV on the same day (co-administration) anytime between 31 August 2022 and 30 January 2023.
- Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years: Participants aged 18-64 years, who were enrolled in the Optum Clinformatics Database and received only COVID-19 vaccine anytime between 31 August 2022 and 30 January 2023.
- Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years: Participants aged 18-64 years, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine and SIV on the same day (co-administration) anytime between 31 August 2022 and 30 January 2023. This arm excluded participants with unknown/other region.
- Group 3a, Model 2: SIV Alone, 18-64 Years: Participants aged 18-64 years, who were enrolled in the Optum Clinformatics Database and received only SIV anytime between 31 August 2022 and 30 January 2023.
Arm/Group | Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years | Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 3a, Model 2: SIV Alone, 18-64 Years
Number analyzed (Participants) | 244900 | 143743 | 244820 | 843412
Participants | 1838 | 705 | 1837 | 12715
Statistical Analysis 1: Comparison: Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years; To account for imbalance in participant characteristics between the vaccine exposure groups, an inverse probability of treatment weights (IPTW) was applied. Analysis performed using IPTW method; Test type: Other; Weighted Hazard Ratio = 1.108, 95% CI 2-sided [1.018 to 1.205]
Statistical Analysis 2: Comparison: Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 3a, Model 2: SIV Alone, 18-64 Years; To account for imbalance in participant characteristics between the vaccine exposure groups, an IPTW was applied. Analysis performed using IPTW method; Test type: Other; Weighted Hazard Ratio = 0.634, 95% CI 2-sided [0.606 to 0.664]

2. Primary Outcome: Number of Participants With All Cause Hospitalization Visits: >=65 Years Old
Description: Hospitalization due to any cause is defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility). To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs SIV alone.
Time Frame: as for outcome 1
Population: All eligible participants whose data were observed in this study. This outcome measure presents reporting arms as planned based on the following: participants >=65 years of age for both models: Model 1 (reporting arms included were co-administration of vaccines on the same day and COVID-19 alone), Model 2 (reporting arms included were co-administration of vaccines on the same day [excluded participants with unknown/other region] and SIV alone).
Measure: Count of Participants; unit: Participants
Groups:
- Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years: Participants aged 65 years and above, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine and SIV (enhanced) on the same day (co-administration) anytime between 31 August 2022 and 30 January 2023.
- Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years: Participants aged 65 years and above, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine anytime between 31 August 2022 and 30 January 2023.
- Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years: Participants aged 65 years and above, who were enrolled in the Optum Clinformatics Database and received COVID-19 vaccine and SIV (enhanced) on the same day (co-administration) anytime between 31 August 2022 and 30 January 2023. This arm excluded participants with unknown/other region.
- Group 3b, Model 2: SIV Alone, >=65 Years: Participants aged 65 years and above, who were enrolled in the Optum Clinformatics Database and received SIV (enhanced) anytime between 31 August 2022 and 30 January 2023.
Arm/Group | Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years | Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 3b, Model 2: SIV Alone, >=65 Years
Number analyzed (Participants) | 382835 | 225680 | 382626 | 1600981
Participants | 7753 | 2719 | 7751 | 33926
Statistical Analysis 1: Comparison: Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.061, 95% CI 2-sided [1.016 to 1.107]
Statistical Analysis 2: Comparison: Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 3b, Model 2: SIV Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 0.897, 95% CI 2-sided [0.875 to 0.919]

3. Primary Outcome: Number of Participants With Composite Coronavirus Disease (COVID-19)-Related Hospitalization, Emergency Department or Urgent Care Visits: Same Day Versus COVID-19 Alone
Description: Hospitalization, emergency department or urgent care visits with COVID-19 diagnosis code (International Classification of Diseases, 10th revision [ICD-10-CM]: U07.1) in any position. To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs SIV alone. In this outcome measure data is reported for Model 1: Same day vs COVID-19 alone.
Time Frame: as for outcome 1
Population: All eligible participants whose data were observed in this retrospective observational study. This outcome measure presents reporting arms as planned based on the following: participants 18-64 years and >=65 years of age for Model 1 (reporting arms included were co-administration of vaccines on the same day and COVID-19 alone).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years | Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years
Number analyzed (Participants) | 244900 | 143743 | 382835 | 225680
Participants | 181 | 55 | 2085 | 684
Statistical Analysis 1: Comparison: Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.543, 95% CI 2-sided [1.133 to 2.1]
Statistical Analysis 2: Comparison: Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.106, 95% CI 2-sided [1.014 to 1.206]

4. Primary Outcome: Number of Participants With Composite Influenza Related Hospitalization, Emergency Department or Urgent Care Visits: Same Day Versus SIV Alone
Description: Hospitalization, emergency department or urgent care visits with Influenza diagnosis code (ICD-10-CM: J09.X, J10.X, J11.X) in any position. To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs SIV alone. In this outcome measure data is reported for Model 2: Same day vs SIV alone.
Time Frame: as for outcome 1
Population: All eligible participants whose data were observed in this retrospective observational study. This outcome measure presents reporting arms as planned based on the following: participants 18-64 years and >=65 years of age for Model 2 (reporting arms included were co-administration of vaccines on the same day [excluded participants with unknown/other region] and SIV alone).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 3a, Model 2: SIV Alone, 18-64 Years | Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 3b, Model 2: SIV Alone, >=65 Years
Number analyzed (Participants) | 244820 | 843412 | 382626 | 1600981
Participants | 145 | 770 | 953 | 3936
Statistical Analysis 1: Comparison: Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 3a, Model 2: SIV Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.048, 95% CI 2-sided [0.903 to 1.217]
Statistical Analysis 2: Comparison: Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 3b, Model 2: SIV Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 0.908, 95% CI 2-sided [0.846 to 0.973]

5. Primary Outcome: Number of Participants With COVID-19 Related Outpatient Visits: Same Day Versus COVID-19 Alone
Description: COVID-19 diagnosis code (ICD-10-CM: U07.1) in any position. An outpatient visit refers to any encounter that is in the outpatient setting. To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs SIV alone. In this outcome measure data is reported for Model 1: Same day vs COVID-19 alone.
Time Frame: From Day 15 of vaccination till end of follow-up observation period, (from 14-Sep-2022 through 14 February 2023 (approximately 5 months); data was extracted and observed in this retrospective study from 05-May-2023 to 12-May-2023 (8 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years | Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years
Number analyzed (Participants) | 244900 | 143743 | 382835 | 225680
Participants | 3513 | 1399 | 6473 | 2268
Statistical Analysis 1: Comparison: Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.137, 95% CI 2-sided [1.068 to 1.211]
Statistical Analysis 2: Comparison: Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.057, 95% CI 2-sided [1.007 to 1.11]

6. Primary Outcome: Number of Participants With Influenza-Related Outpatient Visits: Same Day Versus SIV Alone
Description: Influenza diagnosis code (ICD-10-CM: J09.X, J10.X, J11.X) in any position. An outpatient visit refers to any encounter that is in the outpatient setting. To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs SIV alone. In this outcome measure data is reported for Model 2: Same day vs SIV alone.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 3a, Model 2: SIV Alone, 18-64 Years | Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 3b, Model 2: SIV Alone, >=65 Years
Number analyzed (Participants) | 244820 | 843412 | 382626 | 1600981
Participants | 1346 | 6200 | 1457 | 6396
Statistical Analysis 1: Comparison: Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 3a, Model 2: SIV Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 0.761, 95% CI 2-sided [0.718 to 0.807]
Statistical Analysis 2: Comparison: Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 3b, Model 2: SIV Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 0.858, 95% CI 2-sided [0.811 to 0.907]

7. Primary Outcome: Number of Participants With COVID-19 Related Hospitalization Visits: Same Day Versus COVID-19 Alone
Description: COVID-19 diagnosis code (ICD-10-CM: U07.1) in any position. To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs SIV alone. In this outcome measure data is reported for Model 1: Same day vs COVID-19 alone.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years | Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years
Number analyzed (Participants) | 244900 | 143743 | 382835 | 225680
Participants | 57 | 14 | 452 | 164
Statistical Analysis 1: Comparison: Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.55, 95% CI 2-sided [0.88 to 2.731]
Statistical Analysis 2: Comparison: Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.035, 95% CI 2-sided [0.865 to 1.238]

8. Primary Outcome: Number of Participants With Influenza Related Hospitalization Visits: Same Day Versus SIV Alone
Description: Influenza diagnosis code (ICD-10-CM: J09.X, J10.X, J11.X) in any position. To account for imbalance in participant characteristics between the vaccine exposure groups, 2 separate logistic regression models were used. The two models were: Model 1: Same day vs COVID-19 alone, and Model 2: Same day vs SIV alone. In this outcome measure data is reported for Model 2: Same day vs SIV alone.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 3a, Model 2: SIV Alone, 18-64 Years | Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 3b, Model 2: SIV Alone, >=65 Years
Number analyzed (Participants) | 244820 | 843412 | 382626 | 1600981
Participants | 47 | 228 | 232 | 1164
Statistical Analysis 1: Comparison: Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 3a, Model 2: SIV Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 0.921, 95% CI 2-sided [0.687 to 1.233]
Statistical Analysis 2: Comparison: Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 3b, Model 2: SIV Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 0.826, 95% CI 2-sided [0.722 to 0.945]

9. Primary Outcome: Number of Participants With COVID-19-Related Emergency Department Visits/ Urgent Care Visits: Same Day Versus COVID-19 Alone
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years | Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years
Number analyzed (Participants) | 244900 | 143743 | 382835 | 225680
Participants | 127 | 41 | 1674 | 535
Statistical Analysis 1: Comparison: Group 1a, Model 1: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 2a, Model 1: COVID-19 Vaccine Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.569, 95% CI 2-sided [1.088 to 2.264]
Statistical Analysis 2: Comparison: Group 1b, Model 1: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 2b, Model 1: COVID-19 Vaccine Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.118, 95% CI 2-sided [1.015 to 1.233]

10. Primary Outcome: Number of Participants With Influenza-Related Emergency Department Visits/ Urgent Care Visits: Same Day Versus SIV Alone
Description: as for outcome 8
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years | Group 3a, Model 2: SIV Alone, 18-64 Years | Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years | Group 3b, Model 2: SIV Alone, >=65 Years
Number analyzed (Participants) | 244820 | 843412 | 382626 | 1600981
Participants | 100 | 558 | 736 | 2870
Statistical Analysis 1: Comparison: Group 1a, Model 2: Same Day (COVID-19 Vaccine and SIV), 18-64 Years vs Group 3a, Model 2: SIV Alone, 18-64 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 1.082, 95% CI 2-sided [0.911 to 1.286]
Statistical Analysis 2: Comparison: Group 1b, Model 2: Same Day (COVID-19 Vaccine and SIV), >=65 Years vs Group 3b, Model 2: SIV Alone, >=65 Years; [analysis description as in outcome 1, analysis 2]; Test type: Other; Weighted Hazard Ratio = 0.932, 95% CI 2-sided [0.859 to 1.01]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From Day 1 of vaccination till end of follow-up observation period (approx. 5.5 months, data was extracted and observed in this retrospective study from 05-May-2023 to 12-May-2023 [8 days]); SAEs and Other AEs: Not applicable as safety data not collected.
Description: This observational retrospective study used de-identified data from Optum Clinformatics Database. In this data source, individual identifying information was not available. Minimum criteria for reporting an adverse event could not be met, hence SAEs and other AEs were not planned to be collected and reported.
Arm/Group | Group 1a: Same Day COVID-19 Vaccine and SIV, 18-64 Years | Group 2a: COVID-19 Vaccine Alone, 18-64 Years | Group 3a: SIV Alone, 18-64 Years | Group 1b: Same Day COVID-19 Vaccine and SIV, >= 65 Years | Group 2b: COVID-19 Vaccine Alone, >=65 Years | Group 3b: SIV Alone, >=65 Years
All-Cause Mortality (participants affected / at risk) | 110/244900 | 63/143743 | 794/843860 | 2160/382835 | 1402/225680 | 12031/1601978
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. COVID-19 and influenza vaccinations may have been under-ascertained.
2. The study population included employer-sponsored health plans and Medicare Advantage, which may limit generalizability.
3. It was possible that unmeasured residual confounding remained.
4. Effectiveness for individual influenza vaccines was not assessed.
5. COVID-19 and influenza endpoints were identified using diagnosis codes rather than via laboratory confirmation.
6. This study included only one respiratory virus season.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT05858450/Prot_SAP_000.pdf